CLINICAL TRIAL: NCT03472261
Title: A Randomized Controlled Trial on Integrated Management of Pronation Deformity of Children With Cerebral Palsy Treated by Botulinum Toxin-A
Brief Title: Integrated Management of Pronation Deformity in Cerebral Palsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Nigar Dursun, Professor, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KU GOKAEK 2018/8
Record Dates: First submitted 2018-03-14; First posted 2018-03-21 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; botulinum toxin-A; pronator deformity
MeSH Terms: conditions — Cerebral Palsy | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Patients treated by Botulinum toxin A and twister and specific home exercise program
  Interventions: Drug: Botulinum toxin type A; Other: Upper extremity orthoses; Other: Home exercise program
- Conventional Therapy Group (Active Comparator): Patients treated by Botulinum toxin A and specific home exercise program
  Interventions: Drug: Botulinum toxin type A; Other: Home exercise program

INTERVENTIONS:
Drug: Botulinum toxin type A — Dysport
Other: Upper extremity orthoses — Twister
  Arms: Experimental Group
Other: Home exercise program — Specific exercises for pronation deformity

SUMMARY:
Pronation deformity is a very common problem in children with cerebral palsy. This deformity is usually has neural and non-neural aspects. In this clinical trial the aim is to show the importance of combine treatment approach with pharmacological and non-pharmacological modalities. .

DETAILED DESCRIPTION:
Spasticity is not only the most common motor disorder but also the main cause of slowly developing contractures in children with cerebral palsy. Pronation deformity which is a very common problem in children with cerebral palsy is primarily due to spasticity of the pronator muscles. Reduced strength and loss of control of the supinator muscles and soft tissue and joint contractures usually coexist with spasticity of pronator muscles. There is very limited information about how to treat this deformity in the current literature.

In this prospective, randomized, controlled clinical trial the aim is to show the effectiveness of twister, and home exercise program in an integrated approach with BoNT-A injections on spasticity, and passive range of motion (pROM) of children with CP having pronation deformity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cerebral palsy
* MAS score of pronator muscles at least 2
* Gross Motor Functional Classification Scale level of I-IV
* Scheduled to receive botulinum toxin injections to pronator teres and/or -pronator quadratus muscles besides other spastic upper extremity muscles

Exclusion Criteria:

* Severe cognitive or behavioural problems
* Less than 40 degrees of available passive range of motion in pronation
* Severe dystonia in the affected upper limb
* Received orthopedic surgery to affected upper limb

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline Modified Ashworth Scale (MAS) | Week 12
  Tone measurement

SECONDARY OUTCOMES:
Mean change from baseline passive range of supination | Week 12
  Range of motion measurement
Mean change from baseline angle of catch (XV3) Tardieu scale | Week 12
  Spasticity measurement
Mean change from baseline active range of supination | Week 12
  Active range of motion

OTHER OUTCOMES:
Assisting Hand Assessment (AHA) | Week 12
  Bilateral hand use

CONTACTS AND LOCATIONS:
Overall Officials: Melike Akarsu, MSc, Principal Investigator — Kocaeli University
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)